CLINICAL TRIAL: NCT02127489
Title: The Effects of Single-dose Rectal Midazolam Application on Post-operative Recovery, Sedation, and Analgesia in Children Given Caudal Anesthesia Plus Bupivacaine
Brief Title: The Effects of Single-dose Rectal Midazolam Application on Post-operative Recovery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, SEDAT SAYLAN, Medical Doctor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.KTU.0.01.00.01/372
Record Dates: First submitted 2014-04-18; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Failed Moderate Sedation During Procedure
Keywords: Bupivacaine, caudal, rectal midazolam, children

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam (Active Comparator): 1 mL/kg bupivacaine 0.25%.
  Interventions: Drug: 1 mL/kg bupivacaine 0.25%.
- saline (Placebo Comparator): 5mL rectal saline
  Interventions: Drug: 1 mL/kg bupivacaine 0.25%.

INTERVENTIONS:
Drug: 1 mL/kg bupivacaine 0.25%. — 40 children between 2 and 10 years of ASA I-II were randomized and they received caudal anesthesia under general anesthesia. Patients underwent the application of caudal block in addition with saline and 1 mL/kg bupivacaine 0.25%. In the postoperative period, Group C (n=20) was given 5mL saline and Group M (n=20) was given 0.30 mg/kg rectal midazolam diluted with 5mL saline. Sedation scale and postoperative pain scale (CHIPPS) of the patients were evaluated. The patients were observed for their analgesic need, first analgesic time, and adverse effects for 24 hours.
  Other Names: AstraZeneca Marcaine

SUMMARY:
This study aimed to compare the efficiency of rectal midazolam addition after applying bupivacaine and caudal anesthesia on postoperative analgesia time, the need for additional analgesics, postoperative recovery, sedation, and to find out its adverse effects in children having lower abdominal surgery.

DETAILED DESCRIPTION:
Summary Background: This study aimed to compare the efficiency of rectal midazolam addition after applying bupivacaine and caudal anesthesia on postoperative analgesia time, the need for additional analgesics, postoperative recovery, sedation, and to find out its adverse effects in children having lower abdominal surgery.

Methods: 40 children between 2 and 10 years of American Society of Anesthesiologist (ASA) I-II stages were randomized and applied caudal anesthesia under general anesthesia. Patients were applied caudal block in addition with saline and 1milliliter/kilograms (mL/kg) bupivacaine 0.25%. In the postoperative period, Group C (n=20) was given 5 milliliter (mL) saline and Group M (n=20) was given 0.30 mg/kg rectal midazolam diluted with 5mL saline. Sedation scale and postoperative pain scale (CHIPPS) of the patients were evaluated. The patients were observed for their analgesic need, first analgesic time, and adverse effects for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* children having lower abdominal surgery

Exclusion Criteria:

* Children with significant respiratory system, circulatory system, liver, and kidney function disorder, history of allergy to the drugs to be studied, those who received analgesic medication before the operation, and those for whom caudal anesthesia is contraindicated

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2005-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Sedation scale and postoperative pain scale (CHIPPS) | 24 hours
  Sedation scale and postoperative pain scale (CHIPPS) of the patients were evaluated. The patients were observed for their analgesic need, first analgesic time, and adverse effects for 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: SEDAT SAYLAN, Med. doctor, Principal Investigator — KANUNI EDUCATION AND RESEARCH HOSPITAL, TRABZON ,TURKEY
Locations (1):
- Karadeniz Technical University Faculty of Medicine, Trabzon, Turkey (Türkiye)

REFERENCES:
- [Background] Mahajan R, Batra YK, Grover VK, Kajal J. A comparative study of caudal bupivacaine and midazolam-bupivacaine mixture for post-operative analgesia in children undergoing genitourinary surgery. Int J Clin Pharmacol Ther. 2001 Mar;39(3):116-20. doi: 10.5414/cpp39116. PMID 11396751
- [Background] Breschan C, Schalk HV, Schaumberger F, Likar R. Experience with caudal blocks in children over a period of 3.5 years. Acta Anaesthesiol Scand Suppl. 1996;109:174-6. No abstract available. PMID 8901998
- [Background] Sumpelmann R, Munte S. Postoperative analgesia in infants and children. Curr Opin Anaesthesiol. 2003 Jun;16(3):309-13. doi: 10.1097/00001503-200306000-00011. PMID 17021476
- [Background] Lee HM, Sanders GM. Caudal ropivacaine and ketamine for postoperative analgesia in children. Anaesthesia. 2000 Aug;55(8):806-10. doi: 10.1046/j.1365-2044.2000.01330-2.x. PMID 10947698
- [Background] Silvani P, Camporesi A, Agostino MR, Salvo I. Caudal anesthesia in pediatrics: an update. Minerva Anestesiol. 2006 Jun;72(6):453-9. PMID 16682915
- [Background] Clausen TG, Wolff J, Hansen PB, Larsen F, Rasmussen SN, Dixon JS, Crevoisier C. Pharmacokinetics of midazolam and alpha-hydroxy-midazolam following rectal and intravenous administration. Br J Clin Pharmacol. 1988 Apr;25(4):457-63. doi: 10.1111/j.1365-2125.1988.tb03330.x. PMID 3382589
- [Background] Kanegaye JT, Favela JL, Acosta M, Bank DE. High-dose rectal midazolam for pediatric procedures: a randomized trial of sedative efficacy and agitation. Pediatr Emerg Care. 2003 Oct;19(5):329-36. doi: 10.1097/01.pec.0000092578.40174.85. PMID 14578832
- [Background] McGrath PJ, McAlpine L. Psychologic perspectives on pediatric pain. J Pediatr. 1993 May;122(5 Pt 2):S2-8. doi: 10.1016/s0022-3476(11)80002-8. PMID 8487132
- [Background] Tyler DC, Tu A, Douthit J, Chapman RC. Toward validation of pain measurement tools for children: a pilot study. Pain. 1993 Mar;52(3):301-309. doi: 10.1016/0304-3959(93)90163-J. PMID 8460048
- [Background] Shavit I, Keidan I, Augarten A. The practice of pediatric procedural sedation and analgesia in the emergency department. Eur J Emerg Med. 2006 Oct;13(5):270-5. doi: 10.1097/00063110-200610000-00005. PMID 16969231
- [Background] Roy RC. Choosing general versus regional anesthesia for the elderly. Anesthesiol Clin North Am. 2000 Mar;18(1):91-104, vii. doi: 10.1016/s0889-8537(05)70151-6. PMID 10935002
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Somri M, Gaitini LA, Vaida SJ, Yanovski B, Sabo E, Levy N, Greenberg A, Liscinsky S, Zinder O. Effect of ilioinguinal nerve block on the catecholamine plasma levels in orchidopexy: comparison with caudal epidural block. Paediatr Anaesth. 2002 Nov;12(9):791-7. doi: 10.1046/j.1460-9592.2002.00916.x. PMID 12519139
- [Background] Solak M, Ulusoy H, Sarihan H. Effects of caudal block on cortisol and prolactin responses to postoperative pain in children. Eur J Pediatr Surg. 2000 Aug;10(4):219-23. doi: 10.1055/s-2008-1072362. PMID 11034509
- [Background] Golianu B, Krane EJ, Galloway KS, Yaster M. Pediatric acute pain management. Pediatr Clin North Am. 2000 Jun;47(3):559-87. doi: 10.1016/s0031-3955(05)70226-1. PMID 10835991
- [Background] Martinez-Telleria A, Cano Serrano ME, Martinez-Telleria MJ, Castejon Casado J. [Analysis of regional anesthetic efficacy in pediatric postop pain]. Cir Pediatr. 1997 Jan;10(1):18-20. Spanish. PMID 9131958
- [Background] Da Conceicao MJ, Coelho L. Caudal anaesthesia with 0.375% ropivacaine or 0.375% bupivacaine in paediatric patients. Br J Anaesth. 1998 Apr;80(4):507-8. doi: 10.1093/bja/80.4.507. PMID 9640159
- [Background] Gann DS, Lilly MP. The neuroendocrine response to multiple trauma. World J Surg. 1983 Jan;7(1):101-18. doi: 10.1007/BF01655918. No abstract available. PMID 6301162
- [Background] Kehlet H. The stress response to surgery: release mechanisms and the modifying effect of pain relief. Acta Chir Scand Suppl. 1989;550:22-8. PMID 2652970
- [Background] Reier CE, George JM, Kilman JW. Cortisol and growth hormone response to surgical stress during morphine anesthesia. Anesth Analg. 1973 Nov-Dec;52(6):1003-10. No abstract available. PMID 4357065
- [Derived] Saylan S, Eroglu A, Dohman D. The effects of single-dose rectal midazolam application on postoperative recovery, sedation, and analgesia in children given caudal anesthesia plus bupivacaine. Biomed Res Int. 2014;2014:127548. doi: 10.1155/2014/127548. Epub 2014 May 5. PMID 24883300
- See also: U.S. National Library of Medicine — http://www.ncbi.nlm.nih.gov/pubmed